CLINICAL TRIAL: NCT03889561
Title: Drink Tap: A Multi-Sector Effort to Promote Water Access and Intake in San Francisco Parks to Improve Beverage Intake and Promote Health
Brief Title: Evaluation of the Impact of Water Access and Promotion in Parks on Beverage Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Anisha I Patel, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 43173
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: Water; Parks; Public spaces; Sugar-sweetened beverages
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improved Water Access, Promotion, and SSB taxes (Experimental): Intervention parks will receive installation of water stations, multicultural water promotion campaign, and SSB taxes
  Interventions: Behavioral: Drink Tap
- Control (No Intervention): SSB taxes

INTERVENTIONS:
Behavioral: Drink Tap — The Drink Tap intervention consists of increased access to safe and appealing drinking water, multicultural water promotion, and soda taxes.
  Arms: Improved Water Access, Promotion, and SSB taxes

SUMMARY:
Sugar-sweetened beverages (SSBs) are a major caloric source and the largest source of added sugars in the American diet. While many cities around the country have adopted anti-SSB policies such as soda taxes to reduce SSB intake, there has yet to be any studies to evaluate if the effects of these taxes, coupled with increased water access and promotion effort can lead to decreased sugar sweetened beverage consumption and increased water consumption. This quasi-experimental study evaluates how implementation of SSB taxes, installation of new water stations, and a multicultural water promotion campaign in parks impacts beverage intake in these settings as compared to soda taxes alone.

DETAILED DESCRIPTION:
Consumption of water, in place of sugar sweetened beverages (SSBs), can help prevent obesity and dental carries. While drinking water is associated with these and many other positive health outcomes, many do not meet the recommended dietary intake of water. This is more profound in low income and minority communities that are more likely to drink less water and drink more SSBs. School-based water promotion interventions have shown that improved access to clean drinking water coupled with promotion leads to increases in water consumption and improved health outcomes. No studies have studied the impact of similar strategies on beverage intake and health in parks and public spaces. Parks are an inconspicuous and widely utilized public space, with the majority of Americans going to a park in the last month. This study's central hypothesis is that visitors in parks with SSB taxes coupled with increased access to appealing drinking water and rigorous promotion of its consumption will be more likely to drink water and less likely to drink SSBs, compared to visitors in parks with only SSB taxes. This quasi-experimental study makes use of naturally-occurring policy changes in the San Francisco (SF) Bay Area to disentangle the impacts of anti- SSB policies, water station installation, and multicultural water promotion efforts, using control groups to isolate the effects of anti-SSB policies alone or no intervention. This study will analyze beverage consumption in 10 SF parks that received new water stations and a multicultural water promotion campaign compared to 20 matched control parks (10 parks SF and 10 parks in Oakland) with only SSB taxes.

ELIGIBILITY:
Inclusion Criteria:

* Park visitors within a defined geographic boundary

Exclusion Criteria:

* Park visitors outside a defined geographic boundary

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1038 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in beverage consumption | Visitors in each park will be observed during four one-hour intervals for a maximum of four hours if they visit the park for that duration of time.
  Changes in beverage consumption will be measured through site observations to tally the proportion of visitors drinking water and SSBs in parks.

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Patel, MD,MSPH, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No